CLINICAL TRIAL: NCT00131417
Title: Comparison of the Efficacy of a Ready-to-Use Therapeutic Food With a Milk-Based Diet in the Rehabilitation of Severely Malnourished Ugandan Children
Brief Title: Ready to Use Therapeutic Food in the Rehabilitation of Severely Malnourished Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: NUFU (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002/HD11/244U/RCT
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2005-10-05 (Estimated); Status verified 2005-08

CONDITIONS: Malnutrition
Keywords: severe; malnutrition; ready-to-use-therapeutic-food; children; Uganda
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular

INTERVENTIONS:
Drug: ready-to-use therapeutic food

SUMMARY:
Severe malnutrition is a major cause of child morbidity and mortality in developing countries especially sub-Saharan Africa. The hospital mortality rate due to severe malnutrition in developing countries ranges from 20-30%. For the rehabilitation of severely malnourished children, the World Health Organization (WHO) recommends a liquid milk-based diet, Formula 100 (F100), which contains 100 kilocalories per 100 milliliters. In Uganda, the rehabilitation of severely malnourished children is based on High Energy Milk (HEM), which is reconstituted cows milk with a nutritional composition similar to F100. Recently a semi-solid ready-to-use therapeutic food (RUTF) with similar composition as F100 or HEM has been designed. This preparation can be eaten without adding water hence reducing the risk of bacterial contamination. The preparation can be used at home with minimal supervision. Hitherto the efficacy of RUTF in the rehabilitation of severely malnourished children in Uganda has not been studied. The purpose of this study is to determine whether giving daily RUTF in the rehabilitation of severely malnourished children will result in a higher weight gain than giving HEM.

DETAILED DESCRIPTION:
Severe malnutrition is a major cause of child morbidity and mortality in developing countries especially sub-Saharan Africa. The hospital case fatality rate of severely malnourished children in developing countries ranges from 20 to 30%. In Uganda the prevalence of malnutrition remains high: among children below 5 years, 39% are stunted, 4% are wasted and 23% are under weight. For the rehabilitation of severely malnourished children, the World Health Organization recommends a liquid milk-based diet, formula 100 (F100) which contains 100 kilocalories per 100 milliliters. F100 is prepared by mixing dried skimmed milk, oil, sugar and mineral vitamin mix. It provides 100 kilocalories of energy and contains 2.9 grams of protein per 100 milliliters. In Uganda the rehabilitation of severely malnourished children is based on High Energy Milk (HEM) which is reconstituted cows' milk with nutritional composition similar to F100.

Recently a semi-solid ready- to- use therapeutic food (RUTF) whose nutrition composition is similar to F100 or HEM has been designed. It is prepared by mixing full cream powder, icing sugar, ground nut paste, vegetable oil and mineral vitamin mix. RUTF contains 545 kilocalories per 100 grams of which 10% are protein calories and 59% lipid calories. This preparation can be eaten without adding water hence reducing the risk of bacterial contamination and it can be used at home with minimum supervision. RUTF has energy density of more than 5 times that of milk-based feeds. Hitherto the efficacy of RUTF in the rehabilitation of severely malnourished children in Uganda has not been studied. The purpose of this study is to determine whether giving daily RUTF in the rehabilitation of severely malnourished children results in a higher weight gain than giving HEM.

Hypothesis: Giving 5 meals of RUTF daily in the rehabilitation of severely malnourished children will result in a higher mean weight gain (>10g/kg/day) than giving 5 meals of HEM daily.

The researchers calculated the minimum sample size of 64 patients in each group for 90% power and 95% confidence. In the calculation the researchers assumed that the mean weight gain in the control (HEM) group would be 10.1 g/kg/day with standard deviation of 4.4g according to results of a study by Diop in Senegal; and assumed that the mean weight gain in the RUTF group would be 12.63g/kg/day (25.05% effect size)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 months with severe malnutrition (weight for height less than 70% of median National Center for Health Statistics [NCHS]/WHO reference values)
* Parent's or caretaker's informed consent for study and HIV test.
* Children who have completed initial phase of management of severe malnutrition(without oedema, diarrhoea, vomiting; with normal temperature and gaining weight >5g/kg/day)

Exclusion Criteria:

* Serious medical conditions e.g. severe pneumonia, cerebral palsy
* Persistent diarrhoea

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128
Dates: Start 2004-10; Study Completion 2005-02

PRIMARY OUTCOMES:
mean weight gain (g/kg/day)
time (days) taken to attain 85% weight for height

SECONDARY OUTCOMES:
mortality
adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Nambuya, MBChB, Principal Investigator — Department of Paediatrics and Child Health , Makerere University
Locations (2):
- Centre for International Health University of Bergen, Bergen, Bergen, Norway
- Department of Paediatrics and Child Health, Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Background] Rice AL, Sacco L, Hyder A, Black RE. Malnutrition as an underlying cause of childhood deaths associated with infectious diseases in developing countries. Bull World Health Organ. 2000;78(10):1207-21. PMID 11100616
- [Background] Diop el HI, Dossou NI, Ndour MM, Briend A, Wade S. Comparison of the efficacy of a solid ready-to-use food and a liquid, milk-based diet for the rehabilitation of severely malnourished children: a randomized trial. Am J Clin Nutr. 2003 Aug;78(2):302-7. doi: 10.1093/ajcn/78.2.302. PMID 12885713
- [Background] Ciliberto MA, Sandige H, Ndekha MJ, Ashorn P, Briend A, Ciliberto HM, Manary MJ. Comparison of home-based therapy with ready-to-use therapeutic food with standard therapy in the treatment of malnourished Malawian children: a controlled, clinical effectiveness trial. Am J Clin Nutr. 2005 Apr;81(4):864-70. doi: 10.1093/ajcn/81.4.864. PMID 15817865
- [Background] World Health Organization Mangement of severe malnutrition:a manual for physicians and other health workers, WHO, Geneva. http://www.who.int/nut/documents/manage_severe_malnutrition_eng.pdf (accessed , August, 2004)
- [Background] Briend A, Lacsala R, Prudhon C, Mounier B, Grellety Y, Golden MH. Ready-to-use therapeutic food for treatment of marasmus. Lancet. 1999 May 22;353(9166):1767-8. doi: 10.1016/S0140-6736(99)01078-8. No abstract available. PMID 10347999